CLINICAL TRIAL: NCT07196969
Title: Effects of Electric and Manual Toothbrushes on Periodontal Health and Oral Microbial Flora in Children With Space Maintainers: A Randomized Controlled Trial
Brief Title: Effects of Electric Toothbrushes on Periodontal Health and Oral Microbial Flora in Children With Space Maintainers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Arif Bolaca, Assist. Prof. Dr., Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2022DİŞF002
Record Dates: First submitted 2025-09-21; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Periodontal Parameters; Oral Microbial Colonization; Periodontal Health
Keywords: Electric toothbrush; Manual toothbrush; Periodontal health; Pediatric dentistry; Space maintainers; Salivary microbiota

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group I: Fixed Space Maintainer with Manual Toothbrush (Other): In this group, patients with fixed space maintainers used manual toothbrushes (Oral-B Cavity Defense; Procter & Gamble, USA) during study period.
  Interventions: Device: Manual toothbrush
- Group II: Fixed Space Maintainer with Electric Toothbrush (Experimental): In this group, patients with fixed space maintainers used electric toothbrushes (Oral-B Vitality Cross Action; Procter & Gamble, USA) during study period.
  Interventions: Device: Electric toothbrush
- Group III: Removable Space Maintainer with Manual Toothbrush (Other): In this group, patients with removable space maintainers used manual toothbrushes (Oral-B Cavity Defense; Procter & Gamble, USA) during study period.
  Interventions: Device: Manual toothbrush
- Group IV: Removable Space Maintainer with Electric Toothbrush (Experimental): In this group, patients with removable space maintainers used electric toothbrushes (Oral-B Vitality Cross Action; Procter & Gamble, USA) during study period.
  Interventions: Device: Electric toothbrush

INTERVENTIONS:
Device: Electric toothbrush — Two minutes; twice a day; 3-months.
  Arms: Group II: Fixed Space Maintainer with Electric Toothbrush; Group IV: Removable Space Maintainer with Electric Toothbrush
Device: Manual toothbrush — Two minutes; twice a day; 3-months.
  Arms: Group I: Fixed Space Maintainer with Manual Toothbrush; Group III: Removable Space Maintainer with Manual Toothbrush

SUMMARY:
Objectives: To evaluate and compare the effects of electric and manual toothbrushes on periodontal health parameters and salivary microbial flora in children with fixed and removable space maintainers.

Materials and methods: Sixty-eight children (30 girls, 38 boys; mean age 8.8 years) requiring fixed (n=34) or removable (n=34) space maintainers were randomly allocated to electric (n=17) or manual (n=17) toothbrush subgroups. Periodontal indices; plaque index (PI), gingival index (GI), bleeding on probing (BOP), probing pocket depth (PPD) and salivary levels of Streptococcus mutans and Lactobacillus were assessed at baseline (T0), 1 month (T1), and 3 months (T2).

DETAILED DESCRIPTION:
A total of 68 patients (thirty girls and thirty-eight boys), aged between 6 and 12 years (mean age 8.8), who received either fixed or removable space maintainers due to premature loss of primary molar teeth, were included in the study.

Patients were randomized into two groups based on the type of space maintainer: fixed (n = 34) or removable (n = 34). Each group was further subdivided according to the type of toothbrush used: manual or electric, resulting in four subgroups (n=17). To standardize the study population, only band-and-loop appliances were used in the fixed space maintainer group, which were cemented using a fluoride-releasing glass ionomer cement (RelyX; 3M ESPE, St. Paul, MN, USA). Removable space maintainers consisted of an acrylic base with retention elements such as Adams' clasps, C clasps, or vestibular archesPatients in the removable space maintainer group were instructed to use their appliances during the day, except while eating and sleeping, and to clean them by brushing after toothbrushing.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-12 years who required a space maintainer due to premature loss of primary molar teeth were included if they were medically healthy; had no periodontal disease, temporomandibular disorders, bruxism, abnormal oral habits, or physical/mental disabilities affecting hand movement; were not on regular medication; had not used antibiotics within the past three months or plaque-preventive agents within the last six months; and were able to comply with scheduled follow-up visits.

Exclusion Criteria:

* Patients who failed to attend follow-up appointments or developed an infection/disease requiring antibiotic therapy during the study were excluded.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Change in Plaque Index (PI) | Baseline (T0), 1 month (T1), and 3 months (T2).
  Evaluation of plaque index scores using the Modified Silness and Löe Index.
Change in Gingival Index (GI) | Baseline (T0), 1 month (T1), and 3 months (T2)
  Evaluation of gingival index scores using the Gingival Index.
Change in Bleeding on Probing (BOP) | Baseline (T0), 1 month (T1), and 3 months (T2)
  Evaluation of bleeding on probing scores using the Bleeding on Probing (bop) Index
Change in Periodontal Pocket Depth (PPD) | Baseline (T0), 1 month (T1), and 3 months (T2)
  Evaluation of periodontal pocket depth (PPD)
Change in salivary Streptococcus mutans levels | Baseline (T0), 1 month (T1), and 3 months (T2)
Change in salivary Lactobacillus levels | Baseline (T0), 1 month (T1), and 3 months (T2)

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University Faculty of Dentistry, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No